CLINICAL TRIAL: NCT02237924
Title: Effect of Endostar Combined With Intensity-modulated Radiotherapy Compare With Chemoradiation for Locoregionally Advanced,Low-risk Nasopharyngeal Carcinoma.
Brief Title: Endostar Combined With Intensity-modulated Radiotherapy Compare With Chemoradiation for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, min kang, doctor, First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S201413__19
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; endostar; IMRT; chemoradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endostar + IMRT (Experimental)
  Interventions: Drug: endostar; Radiation: IMRT
- DDP + IMRT (Active Comparator)
  Interventions: Drug: DDP; Radiation: IMRT

INTERVENTIONS:
Drug: endostar — Endostar 7.5mg / m2, 2 cycles of continuous intravenous pumping for ten days,and 2 cycles of maintenance therapy after radiotherapy
  Arms: endostar + IMRT
Drug: DDP — DDP:100mg/m2 for 2-3 cycles
  Arms: DDP + IMRT
Radiation: IMRT — IMRT:70-74Gy for 2-3 cycles

SUMMARY:
A total of 120 patients with pathologically confirmed locally advanced low-risk nasopharyngeal carcinoma were enrolled. They were randomly divided into two groups, with 60 patients in each group. One group was treated with intensity-modulated radiation therapy (IMRT) combined with Endostar and the other group was treated with IMRT combined with concurrent chemotherapy. The short term efficacy and the toxic and side effects of these treatments were evaluated. The 1-year, 3-year, 5-year overall survival and progression-free survival of patients were analyzed. Our data may provide an alternative option for the treatment of locally advanced low-risk nasopharyngeal carcinoma with high efficacy and low toxicity.

DETAILED DESCRIPTION:
This study was a multicenter, open-label, randomized controlled clinical trial. A set of unified standards were used, including the clinical research program, inclusion criteria, exclusion criteria, chemoradiotherapy regimen and evaluation criteria. Nine medical centers participated in this study and 120 patients with pathologically confirmed locally advanced low-risk nasopharyngeal carcinoma were enrolled. These patients were stratified according to clinical stage and participating center, and were randomly divided into two groups: IMRT combined with Endostar group ( IMRT 70-74Gy, Endostar 7.5mg / m2, 2 cycles of continuous intravenous pumping, and 2 cycles of maintenance therapy after radiotherapy) and IMRT combined with concurrent chemotherapy group ( IMRT 70-74Gy, DDP 100mg / m2, intravenous infusion over 2 hours , for 2-3 cycles). After treatment, follow-up was performed every 3 months. The treatment toxicity, local control rate, distant metastasis-free survival, overall survival, progression-free survival were observed and assessed.

ELIGIBILITY:
Inclusion Criteria:

1. patients of either gender and aged from 18 to 70 years old.
2. patients with histologically confirmed non-keratinizing squamous cell nasopharyngeal carcinoma.
3. patients at stage III/IVM0 by UICC2010 staging; patients with higher risk factors (such as N3 and T4N2-phase lymph node ≥4 cm) were excluded.
4. KPS ≥ 70 (Appendix I)
5. patients with available MRI data of nasopharynx and measurable tumor lesions.
6. patients did not receive any treatment before enrollment.
7. patients with expected survival longer than 6 months.
8. biochemical indexes: hemoglobin > 120 g/L, WBC > 4 x 109 /L, and blood platelet ≥ 100 x 109 /L; levels of indicators for hepatic and renal function was 1.25 folds of the upper limit of normal value.
9. the informed content was obtained from every patient.
10. patients with effective follow-up.

Exclusion Criteria:

1. those with malignant tumors other than nasopharyngeal carcinoma, stage I non-melanoma skin cancer, and cervical carcinoma in situ.
2. those received treatments before enrollment.
3. pregnant or lactating women and reproductive women without contraception.
4. those who were undergoing other drug trials.
5. those with severe complications, including myocardial infarction, severe arrhythmia, severe cerebrovascular disease, ulcer disease, mental illness and uncontrollable diabetes.
6. those who could not be followed up at regular intervals.
7. those who were treated with tumor targeting drugs.
8. those who could not subject to MRI examination.
9. those who could not meet the requirements of the prescribed dose.
10. those with hemorrhagic tendency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2021-09 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
5-year Overall Survival | 6 years
  The subjects were randomly divided into two groups. Group A: IMRT combined with Endostar ，including 2 cycles of continuous intravenous pumping, and 2 cycles of maintenance therapy after radiotherapy，and Group B: IMRT combined with concurrent chemotherapy for 2 or 3 cycles. After treatment, the subjects go to observation period for 5 years.

SECONDARY OUTCOMES:
3-year Progression Free Survival | 4 years
  The subjects were randomly divided into two groups. Group A: IMRT combined with Endostar ，including 2 cycles of continuous intravenous pumping, and 2 cycles of maintenance therapy after radiotherapy，and Group B: IMRT combined with concurrent chemotherapy for 2 or 3 cycles. After treatment, the subjects go into observation period. MRI will be used for evaluating the carcinoma status. During 3 years, any relapse or death will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng ren Wang, doctor, Study Director — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Background] Lee AW, Sze WM, Au JS, Leung SF, Leung TW, Chua DT, Zee BC, Law SC, Teo PM, Tung SY, Kwong DL, Lau WH. Treatment results for nasopharyngeal carcinoma in the modern era: the Hong Kong experience. Int J Radiat Oncol Biol Phys. 2005 Mar 15;61(4):1107-16. doi: 10.1016/j.ijrobp.2004.07.702. PMID 15752890
- [Background] Yeh SA, Tang Y, Lui CC, Huang YJ, Huang EY. Treatment outcomes and late complications of 849 patients with nasopharyngeal carcinoma treated with radiotherapy alone. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):672-9. doi: 10.1016/j.ijrobp.2004.11.002. PMID 15936544
- [Background] Yi JL, Gao L, Huang XD, Li SY, Luo JW, Cai WM, Xiao JP, Xu GZ. Nasopharyngeal carcinoma treated by radical radiotherapy alone: Ten-year experience of a single institution. Int J Radiat Oncol Biol Phys. 2006 May 1;65(1):161-8. doi: 10.1016/j.ijrobp.2005.12.003. Epub 2006 Mar 20. PMID 16542792
- [Background] Lee NY, Zhang Q, Pfister DG, Kim J, Garden AS, Mechalakos J, Hu K, Le QT, Colevas AD, Glisson BS, Chan AT, Ang KK. Addition of bevacizumab to standard chemoradiation for locoregionally advanced nasopharyngeal carcinoma (RTOG 0615): a phase 2 multi-institutional trial. Lancet Oncol. 2012 Feb;13(2):172-80. doi: 10.1016/S1470-2045(11)70303-5. Epub 2011 Dec 15. PMID 22178121
- [Background] Pow EH, Kwong DL, McMillan AS, Wong MC, Sham JS, Leung LH, Leung WK. Xerostomia and quality of life after intensity-modulated radiotherapy vs. conventional radiotherapy for early-stage nasopharyngeal carcinoma: initial report on a randomized controlled clinical trial. Int J Radiat Oncol Biol Phys. 2006 Nov 15;66(4):981-91. doi: 10.1016/j.ijrobp.2006.06.013. PMID 17145528
- [Background] Chan AT, Teo PM, Ngan RK, Leung TW, Lau WH, Zee B, Leung SF, Cheung FY, Yeo W, Yiu HH, Yu KH, Chiu KW, Chan DT, Mok T, Yuen KT, Mo F, Lai M, Kwan WH, Choi P, Johnson PJ. Concurrent chemotherapy-radiotherapy compared with radiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: progression-free survival analysis of a phase III randomized trial. J Clin Oncol. 2002 Apr 15;20(8):2038-44. doi: 10.1200/JCO.2002.08.149. PMID 11956263
- [Background] Lee AW, Lau WH, Tung SY, Chua DT, Chappell R, Xu L, Siu L, Sze WM, Leung TW, Sham JS, Ngan RK, Law SC, Yau TK, Au JS, O'Sullivan B, Pang ES, O SK, Au GK, Lau JT; Hong Kong Nasopharyngeal Cancer Study Group. Preliminary results of a randomized study on therapeutic gain by concurrent chemotherapy for regionally-advanced nasopharyngeal carcinoma: NPC-9901 Trial by the Hong Kong Nasopharyngeal Cancer Study Group. J Clin Oncol. 2005 Oct 1;23(28):6966-75. doi: 10.1200/JCO.2004.00.7542. PMID 16192584
- [Background] Wen QL, Meng MB, Yang B, Tu LL, Jia L, Zhou L, Xu Y, Lu Y. Endostar, a recombined humanized endostatin, enhances the radioresponse for human nasopharyngeal carcinoma and human lung adenocarcinoma xenografts in mice. Cancer Sci. 2009 Aug;100(8):1510-9. doi: 10.1111/j.1349-7006.2009.01193.x. Epub 2009 May 21. PMID 19459845